CLINICAL TRIAL: NCT05977335
Title: Continuous and Non-invasive Measurements by Task Force® CORE/CARDIO in Autonomic Function Testing (AFT)
Status: Not yet recruiting | Type: Observational
Sponsor: CNSystems Medizintechnik GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AFTs Task Force® CORE/CARD
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Autonomic Dysfunction; Orthostatic Intolerance
Keywords: Blood Pressure; Hemodynamics; Non-invasive; Continuous; Autonomic Function Testing
MeSH Terms: conditions — Primary Dysautonomias; Orthostatic Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Orthostatic Intolerance Patients
  Interventions: Diagnostic Test: Autonomic Function Testing

INTERVENTIONS:
Diagnostic Test: Autonomic Function Testing — Autonomic Function Testing (AFT) includes Valsalva Manoever, Deep Breathing Test, and Head-up Tilt Table Testing.

SUMMARY:
Background: The investigational device, "Task Force® CORE" (TFC, CNSystems Medizintechnik GmbH, Graz, Austria) together with the "Task Force® CARDIO" (TFCARDIO, CNSystems Medizintechnik GmbH, Graz, Austria) medical device software, is a new CE-marked medical device for continuous non-invasive determination of blood pressure (BP), cardiac output (CO) and derived parameters based on the well established CNAP® (continuous non-invasive arterial pressure) technology by CNSystems.

Aim: The primary aim of this prospective, method comparison, open study is data acquisition for the performance evaluation of the TFC during autonomic function testing in comparison with an clinically accepted reference method. Setting: The setting of the clinical investigation will be the autonomic function testing laboratory at the Department of Neurology, the University Hospital Center Zagreb.

Inclusion criteria: Patients who are over 18 years and who provide written informed consent.

Sample size: The study has an calculated sample size of 70 patients. Considering a drop-out rate of 5%, a total of 75 patients will be included.

Statistics: Descriptive statistics, values for the percentage error and correlation estimates will be derived. Furthermore, scatterplot, Bland-Altman analysis, concordance analysis of parameter changes and further comparative statistics will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (patients aged ≥ 18 years)
* Patients giving written informed consent to participate in the study.
* Patients with intact perfusion of both hands evidenced by a positive Allen's test.
* Patients with orthostatic intolerance will be included

Exclusion Criteria:

* Patients with vascular implants at the sites of non-invasive BP measurement (fingers or upper arms)
* Very low perfusion in the periphery
* Arterial vascular diseases (arteriosclerosis, Raynaud's syndrome, endarteritis obliterans, collagenosis, severely advanced vascular diseases (PAOD))
* Patients with significant edema in the fingers
* Patients with atrial fibrillation
* Patients with valvular disease of grade 2 or above
* Patients with ventricular assist devices
* Subjects not passing the Allen's test for both hands.
* Patients with a large lateral difference in BP (> 15 mmHg for systolic BP and/or >10 mmHg for diastolic BP) or with same arm measurement differences > 10 mmHg in systolic or diastolic BP during assessment of lateral differences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present at the Referral Center for Autonomic Nervous System of the University Hospital Center Zagreb referred to autonomous nervous system testing will be included.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Agreement of blood pressure between investigational and reference device. | The agreement is calculated for the 5 minutes supine baseline period
  The agreement of blood pressure variables [systolic, diastolic and mean pressure in mmHg [millimetres of mercury)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of blood pressure between investigational and reference device. | The agreement is calculated for 60 seconds: during (15 seconds) plus after (45 seconds) valsava maneuver
  The agreement of blood pressure variables [systolic, diastolic and mean pressure in mmHg [millimetres of mercury)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of blood pressure between investigational and reference device. | The agreement is calculated for 90 seconds Deep Breathing period
  The agreement of blood pressure variables [systolic, diastolic and mean pressure in mmHg [millimetres of mercury)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of blood pressure between investigational and reference device. | The agreement is calculated for 10 minutes head-up tilt table test period
  The agreement of blood pressure variables [systolic, diastolic and mean pressure in mmHg [millimetres of mercury)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of heart rate between investigational and reference device. | The agreement is calculated for the 5 minutes supine baseline period
  The agreement of heart rate (bpm [beats per minute)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of heart rate between investigational and reference device. | The agreement is calculated for 60 seconds: during (15 seconds) plus after (45 seconds) valsava maneuver
  The agreement of heart rate (bpm [beats per minute)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of heart rate between investigational and reference device. | The agreement is calculated for 90 seconds Deep Breathing period
  The agreement of heart rate (bpm [beats per minute)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of heart rate between investigational and reference device. | The agreement is calculated for 10 minutes head-up tilt table test period
  The agreement of heart rate (bpm [beats per minute)] between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of cardiac output between investigational and reference device. | The agreement is calculated for the 5 minutes supine baseline period
  The agreement of cardiac output (in l/min) between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of cardiac output between investigational and reference device. | The agreement is calculated for 60 seconds: during (15 seconds) plus after (45 seconds) valsava maneuver
  The agreement of cardiac output (in l/min) between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of cardiac output between investigational and reference device. | The agreement is calculated for 90 seconds Deep Breathing period
  The agreement of cardiac output (in l/min) between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.
Agreement of cardiac output between investigational and reference device. | The agreement is calculated for 10 minutes head-up tilt table test period
  The agreement of cardiac output (in l/min) between both devices will be assessed by means of Scatterplot and Bland-Altman analysis.